CLINICAL TRIAL: NCT01870674
Title: A Randomized, Double-blind, Placebo/Active-controlled, Single/Multiple Dose Phase 1 Clinical Study to Investigate the Safety/Tolerability and PK/PD of YH12852 After Oral Administration in Healthy Subjects
Brief Title: Safety/Tolerability and Pharmacokinetics/Pharmacodynamics of YH12852 After Oral Administration in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: YH12852-101
Record Dates: First submitted 2013-05-20; First posted 2013-06-06 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: safety; tolerability; pharmacokinetics; pharmacodynamics
MeSH Terms: interventions — YH12852; prucalopride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- YH12852 (Experimental): <SAD cohort>
  * Experimental: YH12852 1mg/single dose, qd
  * Experimental: YH12852 3mg/single dose, qd
  * Experimental: YH12852 10mg/single dose, qd
  <FSD cohort>
  * Experimental: YH12852 0.5mg/single dose, qd
  * Experimental: YH12852 1mg/single dose, qd
  * Experimental: YH12852 2mg/single dose, qd
  * Experimental: YH12852 3mg/single dose, qd
  <MAD cohort>
  * Experimental: YH12852 0.5mg/repeat dose, qd
  * Experimental: YH12852 1mg/repeat dose, qd
  * Experimental: YH12852 2mg/repeat dose, qd
  * Experimental: YH12852 3mg/repeat dose, qd
    * Each dosing group(except MAD cohort 0.5mg which has single treatment arm taking YH12852 only) contains 12 subjects. 12 subjects are administered YH12852 or placebo/active comparators.(YH12852:placebo:active=8:2:2)
  Interventions: Drug: YH12852
- Prucalopride (Active Comparator): <each cohort> Prucalopride succinate 1.321mg
  Interventions: Drug: Prucalopride
- Placebo (Placebo Comparator): <each cohort> Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YH12852
  Arms: YH12852
Drug: Prucalopride
  Arms: Prucalopride
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to evaluate the safety/tolerability and pharmacokinetics/pharmacodynamics(PK/PD)of YH12852 after oral administration in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* healthy male/female aged 19 to 45 with body mass index(BMI) between 18 and 25kg/m2
* Subject who has no congenital, chronic disease and disease symptoms in medical examination result
* Subject who is judged to be eligible by principal investigator or sub-investigator according to various reasons including their abnormal test results(clinical laboratory test, 12-lead ECG etc)
* Subjects who has signed a written informed consent voluntarily,prior to any procedure, using a form that is approved by the local Institutional Review Board after detail explanation of the purpose, contents, and characteristic of the drug

Exclusion Criteria:

* Subject who has history or presence of clinically significant diseases in liver, kidney, gastrointestinal tract, nervous system, respiratory system, endocrine system, blood tumor, cardiovascular, urinary system, and mental disorder
* Subject who is hypersensitive to components contained in YH12852 or prucalopride or aspirin/antibiotics like drugs
* Medical history of gastrointestinal disease or acid restraining surgery, gastric/ esophagus surgery(excluding appendectomy, hernia surgery)
* Clinically significant abnormal values in diagnostic check within 28 days before the treatment(>1.25 fold of normal upper limit in the levels of AST or ALT, >1.5 fold of normal upper limit in the levels of Total bilirubin, < 80ml/min of Cockcroft-Gault used creatinine clearance
* Subject has over QTc interval of 550 ms or PR interval of 210 ms or QRS interval of 120 ms or QT interval of 500 ms on baseline 12-lead ECG, as determined by the Investigator
* Subject who had taken usual dose of any prescription drugs within 14 days before the treatment or who had used usual dose of OTC drugs within 7 days before the treatment
* Subject who participated in another clinical trail within 2 months before enrolling in this study
* subject who donated whole blood within 2 months or component blood within 1 month before the treatment
* Medically unacceptable contraception used during the clinical trial
* Subject who drank over 30g/day or were detected alcohol positive on test
* Subject who stopped smoking within 3 months before the treatment or weren't able to stop smoking during the hospitalization
* Subject who had a beverage containing caffeine during the hospitalization
* Subjects with clinically significant observations considered as unsuitable based on medical judgment by investigators

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2013-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
the number of adverse events, seriousness of adverse event | D1~Post study visit
significant changes in vital sign | D1~Post study visit
significant changes in 12-lead electrocardiography | D1~Post study visit
significant changes in laboratory test | D1~Post study visit
significant physical exam | D1~Post study visit

SECONDARY OUTCOMES:
Cmax | 0~48 hrs(SAD,FSD cohorts), 0~24 hrs/D5,6 0hr/D7 0~48hrs(MAD cohort)
AUC | 0~48 hrs(SAD,FSD cohorts), 0~24 hrs/D5,6 0hr/D7 0~48hrs(MAD cohort)
Ae | 0~48 hrs(SAD cohort), 0~24 hrs/D7 0~48hrs(MAD cohort)
BSFS | D1~7(SAD, FSD cohorts), D1~14(MAD cohort)
  pharmacodynamics
Frequency of defecation | D1~7(SAD, FSD cohorts), D1~14(MAD cohort)
  pharmacodynamics

CONTACTS AND LOCATIONS:
Locations (1):
- Inje Busan Paik hospital, Busan, South Korea